CLINICAL TRIAL: NCT04652596
Title: Comparative Effectiveness of Two Interventions to Reduce Food Insecurity During the COVID-19 Pandemic
Brief Title: Reducing Food Insecurity During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency); Krupp Family Foundation (Unknown); Waldron Charitable Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-41052; 6007145 (Other Grant/Funding Number: United States Department of Agriculture (USDA)); AD-1603-34662 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2020-11-30; First posted 2020-12-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Food Insecurity
Keywords: Produce prescription program; Mobile markets; Grocery store gift cards; Fruit and vegetable consumption; Low-income families; Social determinants of health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh Connect Produce Prescription Program (Active Comparator): Investigators will partner with a community organization, About Fresh, that administers a produce prescription program (PPR) and operates mobile fresh foods markets. Participants randomized to this comparator will receive a stipend to Fresh Connect PPR to purchase fresh food items available at mobile markets and at independent farmers markets throughout Boston.
  Interventions: Other: Produce prescription program
- Grocery store gift cards (Active Comparator): Participants randomized to this comparator will receive grocery gift cards redeemable at conventional grocery stores.
  Interventions: Other: Grocery store gift cards

INTERVENTIONS:
Other: Produce prescription program — A monthly $150 stipend will be provided to participants for 6 consecutive months to purchase fresh food items at mobile markets and independent farmers markets across Boston.
  Other Names: Fresh Connect
  Arms: Fresh Connect Produce Prescription Program
Other: Grocery store gift cards — A monthly value of $150 in grocery store gift cards redeemable at conventional grocery stores will be provided to participants for 6 consecutive months.
  Arms: Grocery store gift cards

SUMMARY:
This study aims to compare the effectiveness of two interventions to address food insecurity among low-income families with young children during the COVID pandemic. The investigators will conduct a parallel group, randomized controlled trial of 250 families. The first randomly assigned comparator is Fresh Connect, a produce prescription program that provides a stipend for participants to purchase fresh food items at mobile markets and independent farmers markets across Boston. The second comparator is grocery store gift cards, redeemable at conventional grocery stores. In each comparator, participants will be given the equivalent of $150 on a monthly basis for six consecutive months. All participants will be followed for 12 months to assess outcomes that involve food insecurity (primary), fruit and vegetable consumption, healthcare utilization, social service utilization, and physical/emotional health.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child 0-18 months of age
* Child receives care at Boston Medical Center

Exclusion Criteria:

* Planning to move residence outside of Boston within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Food Security | Baseline, monthly for 12-months post-enrollment
  Self-reported food security status measured by USDA validated 18-question food insecurity screening tool with a 30-day lookback period. Responses are scored with total scores corresponding to four categories: high food security, marginal food security, low food security, and very low food security

SECONDARY OUTCOMES:
Change in fruit & vegetable consumption | Baseline, monthly for 12 months post-enrollment
  Self-reported consumption frequency of fruits, fruit juices, and vegetables in the past 30 days measured by 10-item Dietary Screener Questionnaire scale. Each item is scored from "never" to "6 or more times per day". Scoring algorithms convert frequency responses to cup equivalent estimates of average daily dietary intake for fruits and vegetables, using an age and gender coefficient. The higher the score the more daily dietary intake for fruits and vegetables.
Depression Symptoms | Baseline, monthly for 12-months post-enrollment
  Assessed by the Quick Inventory of Depressive Symptoms (QIDS SR-16). This scale is a 16-item self-report measure of depressive symptoms over the past 7 days. Each item is scored 0-3 (0 = no presence of the symptom; 3 = high burden of the symptom), yielding a total score range of 0 to 27. Because of its wide scoring range, the QIDS can be used to detect depressive illness in populations with low symptoms. Lower scores reflect less depressive symptoms.
Symptom Relief | Baseline, monthly for 12-months post-enrollment
  Assessed by the Beck Anxiety Inventory (BAI). This scale is a 21-item self-report measure the severity of self-reported anxiety. Each item is scored 0-3 (0 = not at all; 3 = severely - it bothered me a lot), yielding a total score range of 0 to 63. The lower the score the less self-reported anxiety.
Changes of behavioral activation for depression | Baseline, every 6 months during 12 month post-enrollment
  Assessed by the Behavioral Activation for Depression Scale (BADS). This 25-item self-reported measure is used to track changes weekly in the behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation. The BADS subscales include activation, avoidance/rumination, work/school impairment, and social impairment. Each item is scored 0-6 (0=not at all; 6=completely), yielding a total score range of 0 to 150. High scores indicate greater levels of activation. For all the subscores, high scores are consistent with the subscale name.
Perceived Stress | Baseline, every 6 months during 12 month post-enrollment
  Assessed by Perceived Stress Scale (PSS). This 14-item psychological instrument measures the perception of stress and the degree to which situations in one's life are appraised as stressful. Each item is scored 0-4 (0=never; 4= very often). The scores is obtained by first reversing the scores on items 4, 5, 6, 7, 9, 10, and 13 and then summing the reverse coded items with the rest of the items. The scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Social Support | Baseline, every 6 months during 12 month post-enrollment
  Assessed by Social Adjustment Scale Self-Report (SAS-SR). This 54-item measure examines social and role functioning in six areas: work; social activities; relationships with family; spouse or partner; parent; member of family unit. Items are rated on a 5-point scale. Seven mean scores are generated, six-role areas and one overall means. The mean scores are converted into standard T-scores on the SAS-SR Profile Form. Higher scores indicate greater impairment of functioning.
Medical outcomes social support | Baseline, every 6 months during 12 month post-enrollment
  Assessed by Medical Outcomes Survey Social Support (MOSSS). This 18-item tool comprises 4 functional support scales (emotional/informational, tangible, affectionate, and positive interaction) and an overall social support index. Each item is scored 0-5 (0=none of the time; 5=all of the time). The higher the overall social support index the more support.
Mastery Control | Baseline, every 6 months during 12 month post-enrollment
  Assessed by Pearlin Mastery Scale (PMS). This 7-item tool measures the extent to which an individual regards their life chances as being under their personal control rather than fatalistically ruled. Each item is scored 1-4 (1=strongly agree; 4=strongly disagree) and the values are added. The scores can range from 7 to 28 with higher scores reflect greater mastery.
Self-Esteem | Baseline, every 6 months during 12 month post-enrollment
  Assessed by Rosenberg's Self-Esteem Scale (RSES). This 10-item self-report likert scale evaluates an individual's self-esteem. Each item is scored from strong agree to strongly disagree. The higher the sum of the scores, the higher the self-esteem.
Unmet needs | Baseline, every 3 months during 12 month post-enrollment
  Assessed by WE CARE. This 12-question screening tool assesses needs in 6 domains: parental educational attainment, employment, child care, risk of homelessness, food security, and household heat and electricity. Individuals respond with "Yes", "No", or "Maybe later". Those with unmet needs are provided with a locally developed community resource information sheet.
Self-Reported Food Assistance Program Participation | Baseline, every 6 months during 12 month post-enrollment
  Self-reported participation in food assistance programs including Electronic Benefits Transfer (EBT), Food Stamps/Supplemental Nutrition Assistance Program (SNAP).
Change in Self-Reported Health Status | Baseline, monthly for 12-months post-enrollment
  Self-reported health status measured by a report of health status as excellent, very good, good, fair, or poor and measured by 3-item CDC Healthy Days module for a disarticulation of physical and mental health.
Maternal attitudes and safe infant care practices | Baseline, every 6 months during 12 month post-enrollment
  Assessed by the Pregnancy Risk Assessment Monitoring System (PRAMS). The survey Identifies groups of women and infants at high risk for health problems, monitors changes in health status, and measures progress towards goals in improving the health of mothers and infants.
Impact of COVID-19 | Baseline, every 3 months during 12 month post-enrollment
  The Epidemic - Pandemic Impacts Inventory (EPII) + 4-item self-report of the impact of the pandemic on financial capacity and food purchasing/acquisition patterns. The EPII is newly developed, thus, scoring procedures will be determined by future research.
Program Experience | 6 months post-enrollment, 12 months post-enrollment
  Assessed by 4-item USDA program experience questions. The questions ask about firm type use, dose of program usage, health education, and program satisfaction.
Change in adult acute healthcare utilization | Baseline, every 6 months during 12 month post-enrollment
  Claims data composite measure (all cause hospital admissions and ED visits; Total number of all-cause ED visits; Total number of all-cause discharges from IP).
Total adult patient-level cost of care | Baseline, every 6 months during 12 month post-enrollment
  Measured via claims data
Child healthcare utilization | Baseline, every 6 months during 12 month post-enrollment
  EPIC chart abstractions (number of office visits, hospitalizations, missed appointments, immunization rates)
Child weight | Baseline, every 6 months during 12 month post-enrollment
  EPIC chart abstractions (weight for age)
Child height | Baseline, every 6 months during 12 month post-enrollment
  EPIC chart abstractions (height for age)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey A Egan, MD MSc, Principal Investigator — Boston Medical Center Department of Pediatrics
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04652596/ICF_000.pdf